CLINICAL TRIAL: NCT06674837
Title: Diagnostics and Surveillance of Acute Meningo-encephalitis Among Children in Cambodia With a Focus on Japanese Encephalitis Virus
Acronym: DEMELE-JEV
Status: Not yet recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS0629s
Record Dates: First submitted 2024-10-28; First posted 2024-11-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Japanese Encephalitis
Keywords: Japanese encephalitis; arbovirus
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples and cerebrospinal fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DEMELE-JEV Cohort 1: This group will include children aged 2-14 years who present at the hospital for reasons other than infectious disease suspicion. During the study of the project, 2000 children will be recruited at each study site. All these children will be followed up at one year and two years post-inclusion
- DEMELE-JEV Cohort 2: This group will include children aged 2-14 years who are hospitalized with febrile neurological syndrome (FNS)

SUMMARY:
The primary objective of this study is to quantify the clinical burden of Japanese Encephalitis (JE) and the asymptomatic circulation of JEV among Cambodian children, through two pediatric cohorts: non-febrile children at recruitment and children hospitalized with febrile neurological syndrome (FNS). Secondary objectives include estimating anti-JEV seropositivity rates, identifying individual risk factors and living conditions associated with JEV infection, characterizing clinical and biological profiles related to disease severity, and evaluating the role of deficiencies in interferon (IFN) response in severe JEV infections.

DETAILED DESCRIPTION:
This is an observational prospective study (with cross-sectional and longitudinal designs) involving two pediatric cohorts recruited from Kantha Bopha hospitals in Phnom Penh and Siem Reap. Group 1 will consist of 2000 non-febrile children aged 2-14 years, recruited from trauma units and followed up for two years to monitor JEV seroconversion. Group 2 will include 2000 children hospitalized with FNS, confirmed JE participants will be followed up for one year to assess the severity of JEV infection. Diagnostic tools such as the QIAstat molecular diagnostic platform and ELISA will be used to detect multiple pathogens, including JEV and dengue virus (DENV). Data collection will involve clinical assessments, etiological testing, and environmental surveys. All collected information will be integrated into a centralized database for analysis.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* All children aged between 2 and 14 years.
* No fever or history of fever in the past 14 days.
* Consenting to return to the hospital for follow-up visits.
* Consenting to blood sampling.
* Written informed assent/consent to participate in the study.

Cohort 2

* Hospitalized patients aged between 2 and 14 years.
* Any neurological disorder.
* Any fever within the past 72 hours.
* Written informed assent/consent to participate in the study.
* No contraindication for lumbar puncture (LP).

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: see eligibility
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To quantify Japanese Encephalitis Virus seroconversion in a cohort of asymptomatic children aged 2-14 years | 24 months
  Japanese Encephalitis Virus seroconversion will be determined based on PCR positivity or ELISA results, with confirmatory testing by virus neutralization assays.
  Unit of Measure: Binary measure (presence or absence) of JEV antibodies or presence of JEV RNA

SECONDARY OUTCOMES:
To assess factors related to the clinical severity of JEV infection among children hospitalized with febrile neurological symptoms (FNS) who are confirmed JEV cases. | 12 months
  Severity will be evaluated based on the following clinical indicators:
  * Length of hospital stay (measured in days).
  * Presence of neurological sequelae (binary outcome: presence or absence).
  * Mortality (binary outcome: survival or death). Unit of Measure: Days for hospitalization length; binary measures for sequelae and mortality.

IPD SHARING:
Plan to Share IPD: Undecided
Cambdodia local reglementation will decide de IPD